CLINICAL TRIAL: NCT01209572
Title: Modelling of 24h Energy Expenditure From Heart Rate, Actimetry and Other Parameters Recorded Under Free-living Conditions
Brief Title: Modelling of Energy Expenditure From Heart Rate, Accelerometry and Other Physiological Parameters
Acronym: Modelheart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AU767; IDRCB 2009-A00912-53 (Registry Identifier: Afssaps)
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2010-09

CONDITIONS: Computer Simulation; Energy Expenditure; Energy Metabolism
Keywords: energy expenditure; heart rate; accelerometry; body temperature; heat flow galvanic response of skin
MeSH Terms: interventions — Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- calorimetric chamber (Experimental)
  Interventions: Device: calorimetric chamber
- Free living conditions (Experimental)
  Interventions: Device: Free living conditions

INTERVENTIONS:
Device: calorimetric chamber — Participants stayed 26h in a calorimetric chamber. They performed a series of physical activities such as walking on a treadmill at different speeds, writing, standing, standing-sitting, stepper , rest , sleeping and eating. They also performed a power test on an ergocycle at different speeds.
  Other Names: indirect calorimetry
  Arms: calorimetric chamber
Device: Free living conditions — Volunteers followed the protocol of doubly labeled water to evaluate their energy expenditure during 10 days in free living conditions. For this period, their heart rate, parameters of actimetry and other parameters were recorded.
  Other Names: Doubly labeled water
  Arms: Free living conditions

SUMMARY:
At this time, 24h energy expenditure is rarely assessed under free-living conditions for specific individuals because of the lack of cheap and accurate software/materials to record the energy expenditure. Some affordable and convenient tools (Polar heart rate monitor, Actiheart, SenseWear Armband) are available on the market but the predictive equations comprised into the software provided with these tools generally miscalculate the energy expenditure (by about +/-10%). Because of this deficiency, the investigators have a poor knowledge of the modification of the energy expended during daily life activities and over 24h in subjects belonging to groups of various ages and physiological states. The investigators hypothesise that it could be possible to improve the energy expenditure prediction.

The project aims at providing a mathematical model (equations) that predicts energy expenditure with an error near to 5%. Two groups of 60 sedentary to athletic normal weight volunteers aged between 18-60 years participate to this study. The first group stay for 26h in calorimetric chambers. During this stay energy expenditure ,heart rate, accelerometry, and other parameters are recorded during various activities. These data will serve to construct the model. The same type of recordings are performed on second group of volunteers in free living conditions. Their energy expenditure is measured overall by doubly labeled water. The data of the second group will serve to validate the model. The error percentage of the model is defined by the ratio of the value of the difference between prediction and reference measure to the reference measure. Concordance between predictions and measures will be evaluated by Bland - Altman plots.

DETAILED DESCRIPTION:
All the volunteers have a visit of inclusion in the Centre de Recherche en Nutrition Humaine. During this visit, the volunteers are informed of the methods of the protocol, the taking of samples, the disadvantages and constraints, on the basis of information letter. They have a medical interrogation and a complete clinical examination by an investigatory doctor or Co-investigator. The biological assessment is requiring 10 ml of blood and including: the analysis of the TSH, a blood count, a sedimentation test. Moreover, for the women in age to procreate, the analysis of the beta - HCG is made. To take another blood sample (10 ml) is necessary for the realization of serology HIV/HCV in the volunteers of the group of doubly labeled water, who provide samples of urine and saliva. The results are communicated to the volunteers confidentially.

Following the visit of inclusion and the signature of the consent form, a food consumption survey is performed to evaluate the energy intakes of the volunteers. Moreover, the body composition and the level of physical-activity of the volunteers are evaluated by biphotonic absorptiometry (DEXA) and using questionnaire MAQ (Modifiable Activity Questionnaire, translated and adapted by Vuillemin and Al, 1999), respectively.

The volunteers of the first group (60) performed a maximal aerobic power test on ergocycle to evaluate their maximum aerobic physical capacity (VO2max), in a hospital laboratory. A measurement of the body composition by biphotonic absorptiometry is also carried out to determine their lean and fat mass. Then, the volunteers stay 26 hours in calorimetric rooms (one evening, one night and a day). The data of indirect calorimetry (O2 consumption and production of CO2), heart rate , actimetry and other parameters are taken into account as from midnight. After one night of sleep, the individuals have to carry out series of state or exercises simulating the daily physical-activities (sleeping, writing 15 min, standing-sitting 5 min, standing 15 min, strolling 15 min, rest 20 min, eating 20 min, household 20 min, stepper 20 min, walking on treadmill at increasing speed 3 km/h, 4 km/h, 5 km/h and 6 km/h during 20 minutes). The volunteers have also to answer questionnaires on their perception of hunger, their emotional state and their visual appreciation of 6 food products at 5 times of the day (before and after the breakfast, before and after the lunch and about 16:30 pm). The rest of the time, their activities are free (watching TV, reading, listening radio …). Measurements finish towards 18:00 and volunteers go home. The meals are balanced in proteins/glucides/lipids and cover energy needs. The menus are established by the dieticians. The meals in calorimetric room are prepared in double weighing to make it possible to calculate the actual quantities.

The second group of volunteers (60) follow the protocol of doubly labeled water to evaluate their energy expenditure during 10 days in free living conditions. For this period, their heart rate, parameters of actimetry and other parameters are recorded . The participants of this second group also answer the questionnaires of perception of hunger, emotional state and visual appreciation of 6 food products, over one day at home. The physical data recorded on this second group will be introduced into the predictive equations. The estimated energy expenditure will be compared with the energy expenditure measured by the technique of doubly labeled water. The answers to the questionnaires filled out by the volunteers of the two groups will be also compared.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age: 18-60 years
* BMI between 19 and 25 kg/m²
* subject considered as healthy after clinical examination and medical questionnaire
* subject giving his/her written informed consent
* subject willing to comply with study procedures
* affiliated to National Health Insurance

Exclusion Criteria:

* biological results judged abnormal by investigator
* positive serologies to HIV or HCV
* respiratory failure or cardiovascular problem
* taking medicine : beta blockers, corticoids, anti-inflammatory drug, thyroid hormones, insulin
* abnormal ECG
* more than 10% of weight or gain loss in the three last months
* tumoral, inflammatory, pulmonary, renal, digestive or liver diseases
* surgery made less than 6 months before the study beginning
* thyroid disease
* pregnant women and nursing mother
* insanity
* smoker
* claustrophobic
* no affiliated to national health insurance people
* refusal to sign informed consent
* refusal to be registered on the national volunteers data file
* currently participating or who having got 4500€ in this year before to have participated in another clinical trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
energy expenditure | one point recorded each minute for 26 hours
  indirect calorimetry

SECONDARY OUTCOMES:
energy expenditure | one point at the end of the 10-day period
  doubly labeled water
heart rate | one point recorded each minute for 26 hours or 10 days
  measurements made by electrocardiogram
Accelerometry | one point by minute for 26 hours or 10 days
  uniaxial and biaxial measurements
hunger and emotional state perception | evaluation before and after each meal
  validated questionnaires (Hunger and brief mood introspective scale)
hedonic evaluation of 6 food products | before and after each meal
  home made questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, MD-PhD, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre de Recherche en Nutrition Humaine d'Auvergne, Clermont-Ferrand, Auvergne, France

REFERENCES:
- See also: research fields of the Institute — http://www.inra.fr
- See also: Research fields of CRNH — http://www1.clermont.inra.fr/crnh